CLINICAL TRIAL: NCT02813707
Title: A Prospective Study to Determine Long Term Impact of Bariatric Surgery on Metabolic, Nutritional and Quality of Life Status: PART 2
Brief Title: Prospective Study to Determine Long Term Impact of Bariatric Surgery
Acronym: BS-PART2
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: United Arab Emirates University (Other)
Responsible Party: Principal Investigator, Juma Alkaabi, Professor of Medicine, Consultant Endocrinologist, United Arab Emirates University
Other Study IDs: 16/008 2016 4272
Record Dates: First submitted 2016-05-03; First posted 2016-06-27 (Estimated); Last update posted 2016-06-28 (Estimated); Status verified 2016-06

CONDITIONS: Quality of Life
Keywords: Vitamins; Mineral; Surgery
MeSH Terms: conditions — Calcinosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: QoL questionnaire regarding the long term complication — Micronutrients evaluation

SUMMARY:
The World Health Organization (WHO) statistics, in 2008, there were more than 1.4 billion adults, aged 20 and older, and were overweight. Of these over 200 million men and nearly 300 million women are obese. Body Mass Index (BMI) more than 30 is considered as obese and increasingly bariatric surgery is the commonest way used nowadays to lose weight. Moreover, surgery will influence many other health factors and parameters. Many studies prove the improvement of metabolic and psychological status of patients post bariatric surgery. In addition, many vitamins will be affected and should be replaced. This research study is continuation (PART 2) of previously approved study (approval: 13/54). Brief findings of the study are attached. Our aim in this part of the study to assess long term the impact of bariatric surgery on metabolic, nutritional and quality of life status on patients post bariatric procedure of at least 12 months post-surgery follow up. As we noted in our previous initial study that there is significant loss the collection of the data due to "no show" for proper follow up routine care. Previously it was approved to consent patients by phone calls and extract information regarding Quality of Life (QoL) post-surgery. This will be replaced by seeing the patients in the outpatient clinic and providing the necessary information and consent.

DETAILED DESCRIPTION:
There is no data available in the UAE regarding the impact of bariatric surgery on metabolic, nutritional and psychological status of the patient. Therefore, studying that will help the community in establishing a database specific for the country instead of relying on other countries statistics and data.

In 2009, figures from WHO have revealed that 39.9% of women in United Arab Emirates (UAE) are obese which considered the 7th highest proportion in the world. On the other hand, 25.6% of men are obese in UAE which considered the 9th highest proportion in the world.

The search for ideal weight loss operation started more than 50 years ago. First bariatric surgery performed in 1954 by Kremen and his associates which involved the anastomosis of upper and lower intestine that bypasses large amount of absorptive circuit. Mason, Ito et al. developed the Gastric Bypass in 1967, which led to fewer complications than the intestinal bypass. A later improvement, the Roux-en-Y Gastric Bypass, proved technically difficult to perform but led to long-term sustained weight loss, no protein-calorie malabsorption and little vitamin or mineral deficiencies. Many studies and researches are conducting studying the impact of bariatric surgery on different health parameters.

There are many studies regarding the effect of bariatric surgery on diabetic and metabolic parameters. Study of 15 patients with Body Mass Index (BMI) between 30-35 kg/m2 with type II diabetes underwent Roux-En-Y gastric bypass with 1 year follow up. Results that diabetes mellitus remission achieved in 93% of cases with significant drop in blood glucose and HbA1C (p≤ 0.05 & p ≤ 0.001) respectively. Another study, 17 obese patients with type II diabetes mellitus (DM) received the duodenal-jejunal bypass liner followed for 24 weeks. HbA1C improved from 8.4±0.2 to 7.0±0.2% (p≤0.01). A third study regarding the effect of laparoscopic Roux-En-Y gastric bypass (LRYGBP) on (Diabetes mellitus II) DMII for period of 5 years. 1160 patients underwent LRYGBP and 240 (21%) has impaired fasting glucose (IFG) or DMII. Body mass index (BMI) decreased from 50.1 to 34 kg/m2. Hemoglobin A1C (HbA1C) returned to normal levels (83%) or markedly improved (17%) in all patients. Reduction in use of oral anti-DM (80%) and insulin (79%) followed surgical treatment. Furthermore, in other study 52 morbidly obese patients were studied after sleeve gastrectomy. HbA1C changed form 6.0 ± 1.3% to 5.4 ± 0.8% to 5.4 ± 0.8% at 6 and 12 months respectively. Triglyceride decreased from 159± 87 to 116± 41 and 116± 62 mg/dl, while High density lipoprotein (HDL) increased from 46± 12 to 50 ±12 and 56±13 mg/dl at 6 and 12 months. There is a study of 100 obese patients after laparoscopic adjustable gastric banding and the influence on body mass index (BMI), insulin concentration and lipid profile. Results include significant decrease in BMI, normalization of metabolic parameters, with improvement of type II DM, Hypertension (HTN), and sleep apnea.

There is a study about improving renal function 12 months after bariatric surgery. They studied changes in Glomerular Filtration Rate (GFR) before and 1 year after the surgery in 223 severely obese patients. Normal GFR was 90-125 ml/min. They found that GFR increased in patients with previously normal, Chronic kidney disease (CKD) stage II and CKD stage III. Another 12- month prospective study, regarding the effect of bariatric surgery on renal function and systemic inflammation and blood pressure. A total of 34 morbidly obese patients were investigated at baseline, 1 month and 12 months after Roux-En-Y gastric bypass. The results showed a significant decrease in body mass index (BMI), mean arterial pressure, and urinary and serum inflammatory markers (all p≤0.001). There are many studies in the literature regarding improving quality of life (QoL) after bariatric surgery. There was a study in which obese patient's QoL was investigated early and medium-term changes following Roux-en-y gastric bypass.

There was a study regarding the sexual function post bariatric surgery. In a prospective study of 39 men underwent bariatric surgery. Their sexual function was assessed by mean of international index of erectile function (IIEF) before and 1 year after the surgery. In addition to, metabolic and hormonal parameters (like weight, HbA1C, lipoid profile, insulin sensitivity and sex hormones). They found that erectile function score improved from baseline of 54.85 ± 16.59 to 61.21 ± 14 with P ≤ 0.01 and gonadal function including testosterone level(from 256.36 ± 120.98 in baseline to 508.01±161.90 with P ≤0.01 at 1 year.

There are many studies regarding the nutritional deficiency following bypass surgeries. There is a study of long-term nutritional deficiencies and dietary intake after sleeve gastrectomy or Roux-En-Y gastric bypass in a mediterranean population. It was a longitudinal, prospective and observational study in which primary outcomes were changes in energy, macronutrients, and micronutrients intake and weight loss. They found that the mean daily intake of calcium, magnesium, phosphorus, and iron was less than the current recommendations. The most common observed deficiency is 25-hydroxy vitamin D. On the other hand, there are 2 case reports of night blindness and visual impairment caused by vitamin A deficiency after bariatric surgery which considered a significant complication after mal-absorptive bariatric surgery. Moreover, there is a prospective, single-center, observational study regarding nutritional deficiencies following sleeve gastrectomy with a medium follow up of 2 years. From 100 patients were studied, 48% were supplemented with iron, 33% with zinc, 34% with a combination of calcium carbonate + cholecalciferol, 24% with vitamin D, 42% with vitamin B12, and 40% with folic acid. The patients who received only a sleeve gastrectomy had (Excess weight loss % EWL) of 53.6%, 65.8% and 62.6% after 6, 12 and 24 months, respectively.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients who underwent any type of bariatric surgery at Tawam Hospital with at least 12 months duration post-operative

Exclusion Criteria:

* Not willing to participate in the study.
* No show

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be identified from the list of the bariatric surgery done at Tawam hospital.
  The study will be conducted in Tawam Hospital where patients come for their routine bariatric surgery. A written informed consent will be taken from all the patients willing to participate in the study. Patients would be informed about the objectives / goals of the study.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2016-04; Primary Completion 2016-12 (Estimated); Study Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
Postsurgical complications | 1 year
  changes in body weight
Monitor the HbA1c levels | 1 year
  Changes in the HbA1c Levels

SECONDARY OUTCOMES:
Status renal function | 1 year
  occurrence of renal stone
Monitor the Iron levels | 1year
  Changes in Iron level
Monitor the PTH levels | 1year
  changes in the levels of PTH
Monitor the thiamine level | 1 year
  change in level of thiamine
Monitor the vitamins B12 levels | 1year
  changes in Vitamin B12 levels

CONTACTS AND LOCATIONS:
Overall Officials: Salah Gariballa, MD, Study Chair — United Arab Emirates University
Locations (1):
- Faculty of Medicine and Health Sciences UAE University, Al Ain City, AB, United Arab Emirates